CLINICAL TRIAL: NCT02235194
Title: Influence of an Amino Acid and Chromium Containing Table Water on Glucose Response to a Test Meal in Type 2 Diabetes Patients in a Double Blind Cross - Over Design
Brief Title: Effects of an Amino Acid and Chromium-picolinate Containing Drink on Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stoffwechselzentrum Rhein - Pfalz (Other)
Responsible Party: Principal Investigator, Dr. Per Humpert, Privatdozent Dr. Per M. Humpert, Stoffwechselzentrum Rhein - Pfalz
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SWZRP-14-01
Record Dates: First submitted 2014-08-28; First posted 2014-09-09 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes; Prediabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amino Acids, Chromium - Picolinate (Active Comparator): Verum drink containing the dietary supplements is taken with a test meal. INsulin and glucose response is documented for 180 minutes.
  Interventions: Dietary Supplement: Amino Acid and chromium-picolinate containing drink; Dietary Supplement: Placebo Drink
- Placebo Drink (Placebo Comparator): Placebo Drink containing aroma only is taken with a test meal. INsulin and glucose response is documented for 180 minutes.
  Interventions: Dietary Supplement: Amino Acid and chromium-picolinate containing drink; Dietary Supplement: Placebo Drink

INTERVENTIONS:
Dietary Supplement: Amino Acid and chromium-picolinate containing drink — Amino Acid and chromium - picolinate containg water ist taken with a test meal to study efects on glucose and insulin response.
Dietary Supplement: Placebo Drink — Placebo drink ist taken with a test meal to study efects on glucose and insulin response.

SUMMARY:
It has previously been shown in healthy overweight subjects, that table water including a defined amount of amino acids and chromium can decrease the postprandial glucose and insulin response. In this study, the effect of this table water on glucose excursions after a test meal containing a defined amount of available carbohydrates, protein and fat will be studied in patients with early type 2 diabetes or prediabetes according to guidelines that are treated with dietary measures or metformin only. The study will be conducted in a cross -over design, double blinded and placebo controlled including 20 participants. The primary endpoint of the study is the incremental area under the curve for plasma glucose (iAUCgluc) within 180 minutes after ingestion of the meal.

ELIGIBILITY:
Inclusion Criteria:

* Early Type 2 Diabetes (i.e. on Metformin or diet only)
* Prediabetes (i.e. FPG 100-125 mg/dl or IGT 2h PG in OGTT 140-199 mg/dl)
* HbA1c < 7%
* BMI 28,0-39,9 kg/m²

Exclusion Criteria

* Any antidiabetic medication other than metformin
* Psychiatric Disease
* Acute Infections
* Alcohol or drug abuse
* Malignant tumors or hematologic disorders
* Heart failure NYHA III-IV
* Acute coronary syndrome
* Any macrovascular event within previous 3 months
* Chronic kidney disease > Stage 3
* Pregnancy or Lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Area under the curve for Glucose | 0', 15', 30', 60', 90', 120', 150', 180' post test meal
  Area under the curve for glucose will be measured within 180 minutes after a test meal. Blood samples will be drawan at 8 timepoints during 180 minutes after ingestion of the test meal (0', 15', 30', 60', 90', 120', 150', 180').

SECONDARY OUTCOMES:
AUC for insulin | 0', 15', 30', 60', 90', 120', 150', 180' post test meal
  Blood samples will be drawan at 8 timepoints during 180 minutes after ingestion of the test meal (0', 15', 30', 60', 90', 120', 150', 180').
Markers of inflammation | at 0', 15', 30', 60', 90', 120', 150', 180' post test meal
  Blood samples will be drawan at 8 timepoints during 180 minutes after ingestion of the test meal (0', 15', 30', 60', 90', 120', 150', 180'). At these timepoints markers of inflammation will be measured (i.e. hsCRP and others)
markers of lipid metabolism | 0', 15', 30', 60', 90', 120', 150', 180' post test meal
  Triglycerides, VLDL and other parameters of lipid metabolism are planned to be measured within 180 minutes after a test meal at 0', 15', 30', 60', 90', 120', 150', 180'.
Gut peptide hormones | 0', 15', 30', 60', 90', 120', 150', 180' post test meal
  Area under the curve for GLP-1, ghrelin, glucagone and GIP are measured within 180 minutes after the test meal.

CONTACTS AND LOCATIONS:
Locations (1):
- Stoffwechselzentrum Rhein Pfalz, Mannheim, Germany